CLINICAL TRIAL: NCT01722513
Title: Phase 4 Study of Alprostadil Prevent Contrast Induced Nephropathy in Patients Receiving a Cardiac Catheterization
Brief Title: Efficacy and Safety of Alprostadil Prevent Contrast Induced Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, MD FACC, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: NCT20120312
Record Dates: First submitted 2012-11-03; First posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Kidney Diseases; Diabetes Mellitus; Acute Kidney Injury; Kidney Failure, Chronic; Renal Insufficiency
Keywords: Contrast Induced Nephropathy
MeSH Terms: conditions — Kidney Diseases; Diabetes Mellitus; Acute Kidney Injury; Kidney Failure, Chronic; Renal Insufficiency | interventions — Alprostadil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alprostadil, Control (Experimental): Alprostadil interventions: Alprostadil 40 ug + 1cc/kg/hr normal salin 6 hour before and after angiography AND Control interventions:Normal salin 1cc/kg/hr before and after angiography
  Interventions: Drug: Alprostadil ﹠control

INTERVENTIONS:
Drug: Alprostadil ﹠control — control:Normal salin 1cc/kg/hr before and after angiography
  Other Names: Drug: Alprostadil; lipo-alprostadil; Prostaglandin E1; Drug: normal salin

SUMMARY:
The aim of this prospective, randomized, controlled study is to investigate the effect of pretreatment with intravenous Alprostadil on the incidence of CIN in a high-risk population of patients with both type 2 diabetes mellitus (T2DM) and CKD undergoing coronary angiography, and evaluate the influence of such potential benefit on short-term outcome.

DETAILED DESCRIPTION:
The number of cardiac angiography and percutaneous coronary interventions (PCI) has increased steadily in recent years. This has resulted in the increasing incidence of contrast-induced nephropathy (CIN). Major risk factors for CIN include older age, diabetes mellitus (DM), chronic kidney disease (CKD).

The aim of this prospective, randomized, controlled study is to investigate the effect of pretreatment with intravenous Alprostadil on the incidence of CIN in a high-risk population of patients with both type 2 diabetes mellitus (T2DM) and CKD undergoing coronary angiography, and evaluate the influence of such potential benefit on short-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient that underwent coronary angiography
* T2DM
* CKD stages 2 and 3, eGFR 30 to 89ml/min per 1.73m2
* Alprostadil naive, or not on Alprostadil treatment for at least 14 days
* Withdrawal metformin or aminophylline for 48h before angiography

Exclusion Criteria:

* serum Cr. More than 3 mg/dl
* electrolyte and acid-base imbalance
* pulmonary edema
* allergy to Alprostadil

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 72 h
  An absolute increase in SCr >=0.5mg/dL（>=44.2μmmol/L）or a >= 25% increase in SCr from baseline to 72h after the procedure

SECONDARY OUTCOMES:
Secondary Outcome | 30 d
  The composite of hospitalization for aggravated renal function, acute renal failure, dialysis or hemofiltration, aggravated at least 1 class of heart function, acute left ventricular failure or death from all causes.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Wei Xu, MD, FACC, Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital, Tongji University School of Medicine
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Koch JA, Plum J, Grabensee B, Modder U. Prostaglandin E1: a new agent for the prevention of renal dysfunction in high risk patients caused by radiocontrast media? PGE1 Study Group. Nephrol Dial Transplant. 2000 Jan;15(1):43-9. doi: 10.1093/ndt/15.1.43. PMID 10607766